CLINICAL TRIAL: NCT04305444
Title: Phase II Expansion Cohorts Studies of a Novel Triple Combination Therapy, DTRM-555, in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia or Relapsed/Refractory Non-Hodgkin's Lymphomas
Brief Title: Study of a Triple Combination Therapy, DTRM-555, in Patients With R/R CLL or R/R Non-Hodgkin's Lymphomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite the efforts of our dedicated team and initial progress, we were unable to secure the necessary financial resources to continue the study. We appreciate the support and participation of all involved.
Sponsor: Zhejiang DTRM Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTRM-555_001
Record Dates: First submitted 2020-03-06; First posted 2020-03-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Richter's Transformation
Keywords: B-Cell Lymphoma; Diffuse Large B Cell Lymphoma; Everolimus; Follicular Lymphoma; Immunosuppressive Agents; Leukemia; B-Cell Leukemia; Chronic Lymphocytic Leukemia; Lymphatic Diseases; Lymphoma; Malignant Lymphoma; Non-Hodgkin Lymphoma; Lymphoproliferative Disorders; Neoplasms; Tyrosine Protein Kinase; Bruton's Tyrosine Kinase Inhibitor; Pomalidomide
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell; Leukemia; Leukemia, B-Cell; Lymphatic Diseases; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Neoplasms | interventions — DTRMWXHS-12; Everolimus; pomalidomide

STUDY DESIGN:
Intervention Model Description: All patients, regardless of disease-specific cohort, will receive the same dose of DTRM-555. There are two stages to the study, and there is the potential for 120 patients in total (potentially 24 patients in each of the 5 cohorts) to participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Disease-specific cohorts (Experimental): Participants will be administered the oral triple-combination therapy, DTRM-555 (comprised of 200mg of DTRMWXHS-12, 5mg of everolimus and 2mg of pomalidomide), once-daily for 21 consecutive days every 28 days
  Interventions: Drug: DTRM-555

INTERVENTIONS:
Drug: DTRM-555 — Oral once-daily administration
  Other Names: DTRMWXHS-12; everolimus; pomalidomide

SUMMARY:
Targeted drug therapies have greatly improved outcomes for patients with relapsed or refractory (R/R) chronic lymphocytic leukemia (CLL) and non-Hodgkin's lymphoma. However, single drug therapies have limitations, therefore, the current study is evaluating a novel oral combination of targeted drugs as a way of overcoming these limitations. This study will determine the efficacy of the triple combination therapy, DTRM-555, in patients with R/R CLL or R/R non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This study is being conducted in three parts: Phase Ia, Phase Ib and Phase II, disease-specific expansion cohorts. Phase Ia explored escalating doses of a monotherapy of a novel Bruton's Tyrosine Kinase (BTK) inhibitor, DTRMWXHS-12. Phase Ib explored two combination therapies, DTRM-505 (DTRMWXHS-12 and everolimus) and DTRM-555 (DTRMWXHS-12, everolimus and pomalidomide).

The current Phase II study will further examine the investigational triple combination treatment, DTRM-555 for efficacy and safety. The study is being conducted in five disease-specific cohorts: Activated B-Cell (ABC) Diffuse Large B-Cell Lymphoma, Germinal Center B-Cell (GCB) Diffuse Large B-Cell Lymphoma, Richter's Transformation, transformed Follicular Lymphoma, and relapsed or refractory Chronic Lymphocytic Leukemia.

The Primary Objective of the Phase II study is to determine the efficacy of the triple combination therapy, DTRM-555, in the five disease-specific cohorts. The Secondary Objectives are (1) to determine the safety of DTRM-555 in the cohorts and (2) to obtain the pharmacokinetics of DTRM-555 (i.e., DTRMWXHS-12, everolimus and pomalidomide).

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent.
* Patients with a diagnosis of R/R CLL or other B-cell neoplasms (i.e., ABC DLBCL, GCB DLBCL, Richter's transformation and tFL) who have no available approved therapies, or patients with a diagnosis of non-Hodgkin's lymphoma, which has relapsed and/or is refractory to standard therapy.

  a. Patients with R/R CLL must have been exposed to Bruton's tyrosine kinase (BTK) or B-Cell CLL/Lymphoma 2 (BCL2) inhibitor-based therapy in prior lines of therapy but must not have known Cys481 resistance mutation prior to study enrollment.
* Age ≥ 18 years.
* Life expectancy greater than 12 weeks.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Ability to swallow and retain capsules and/or tablets.
* Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, or other organ dysfunctions.
* If the patient consents to an optional tumor biopsy, he/she must have a tumor that can be safely biopsied and undergo a baseline tumor biopsy procedure, or be willing to provide available archival tissue collected within 6 months of signing the Informed Consent Form (ICF), and one post-Cycle 1 treatment biopsy.
* Patients must have at least one target lesion according to Lugano Classification. Patients with R/R CLL are exempt from this requirement.
* Women of child-bearing potential must have a negative serum or urine pregnancy test.
* Women of child-bearing potential must agree to use 2 reliable methods of contraception beginning 4 weeks prior to the initiation of treatment, during therapy, and for at least 4 weeks after the last drug administration.
* Men must agree to use a latex or synthetic condom during sexual contact with a pregnant female or a female of child-bearing potential, for the duration of the study and for at least 4 weeks after the last drug administration, even if they have undergone a successful vasectomy.

Exclusion Criteria:

* Received prior systemic anticancer treatment within the following time frames:

  1. Chemotherapy, immunotherapy, radiotherapy or any other investigational therapy within 21 days prior to starting study treatment.
  2. Targeted therapies within 5 biological half-lives prior to starting study treatment.
* Patients with active infections requiring therapy are not eligible for entry into the study until resolution of the infection; however, patients on prophylactic antibiotics, antifungals or antivirals are eligible for entry into the study.
* Pregnant or lactating individuals.
* Impaired hepatic or renal function as demonstrated by any of the following laboratory values:

  1. Aspartate transaminase (AST) or alanine transaminase (ALT) > 2.5 x upper limit of normal (ULN); for patients with liver involvement, > 5 x ULN
  2. Total bilirubin > 1.5 x ULN (Patients with a history of Gilbert's syndrome may participate if total bilirubin is less than or equal to 3 x ULN and the AST/ALT and alkaline phosphatase meet the protocol-specified levels for eligibility)
  3. Alkaline phosphatase > 2.5 x ULN
  4. Glomerular filtration rate < 50 mL/min, as assessed using the standard methodology at the investigating center (i.e., Cockcroft-Gault), or serum creatinine > 1.5 x ULN
* International normalized ratio (INR) > 1.5 or other evidence of impaired hepatic synthesis function.
* Absolute neutrophil count < 1.0 x 109/L or platelets < 100 x 109/L, unless due to disease-related bone marrow impairment as confirmed by bone marrow biopsy during screening or due to standard of care treatment within 2 months prior to signing of informed consent. Patients with bone marrow impairment will be excluded if their absolute neutrophil count (ANC) is < 0.5 x 109/L and platelets < 50 x 109/L.
* Previous allogeneic bone marrow transplant is restricted, unless transplant was greater than 3 months prior and there is no evidence of acute or chronic graft versus host disease.
* Central nervous system involvement with malignancy.
* Patients who have poorly controlled diabetes mellitus or whose glucose values cannot be controlled with medical treatment.
* Current malignancies of another type, with the exception of adequately treated in situ cervical cancer and basal cell skin cancer, squamous cell carcinoma of the skin or other malignancies with no evidence of disease for 2 years or more.
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Documented or known bleeding disorder.
* Requirement for anticoagulation treatment that increases INR or activated partial thromboplastin time above the normal range (low molecular weight heparin and heparin line flush allowed).
* Patients requiring the use of strong CYP3A4, CYP1A2, or P-gp inhibitors.
* Patients with a significant cardiovascular disease or condition, including:

  1. myocardial infarction within 6 months of study entry,
  2. New York Heart Association Class III or IV heart failure,
  3. uncontrolled dysrhythmias or poorly controlled angina,
  4. history of serious ventricular arrhythmia (ventricular fibrillation or ventricular tachycardia, ≥ 3 beats in a row) and/or risk factors (e.g., heart failure, hypokalemia, or family history of Long QT Syndrome),
  5. baseline prolongation of QT/QTc interval (repeated demonstration of corrected QT interval (QTc) ≥ 450 msec for men and 470 msec for women), and
  6. left ventricular ejection fraction (LVEF) < 45% by multiple gated acquisition (MUGA) and /or echocardiogram (ECHO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Complete Responses (CR) and Partial Responses (PR) with DTRM-555 in the five disease-specific cohorts | 24 months
  Response in lymphoma patients will be assessed according to Lugano 2014 criteria guidelines for response assessment of Hodgkin and non-Hodgkin lymphoma. Response in CLL patients will be assessed according to International Workshop on CLL (iwCLL) 2018 criteria for treatment of CLL.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events (AEs) in the five disease-specific cohorts | 24 months
  Percentage of participants with Treatment-Emergent Adverse Events (AEs)
Overall Response Rate (ORR) with DTRM-555 in the five disease-specific cohorts | 6, 12 and 24 months
  Response in lymphoma patients will be assessed according to Lugano 2014 criteria guidelines for response assessment of Hodgkin and non-Hodgkin lymphoma. Response in CLL patients will be assessed according to iwCLL 2018 criteria for treatment of CLL.
Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine key pharmacokinetic parameters for the three drugs | 24 hours
  Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine Area Under the Curves (AUC)
Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine key pharmacokinetic parameters for the three drugs | 24 hours
  Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine Maximum Observed Plasma or Blood Concentrations (Cmax)
Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine key pharmacokinetic parameters for the three drugs | 24 hours
  Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine the Times to Reach Cmax (tmax)
Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine key pharmacokinetic parameters for the three drugs | 24 hours
  Plasma or blood concentration versus time profiles of DTRMWXHS-12, everolimus and pomalidomide will be evaluated to determine Elimination Half-Lives (t1/2)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Mayo Clinic, Phoenix, Arizona
  - Yale - Smillow Cancer Hospital, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - VA Medical Center - Memphis, Memphis, Tennessee